CLINICAL TRIAL: NCT04887272
Title: Weathering the Storm: Lung, Heart, and Brain Vascular Rehabilitation for COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Kurt Smith, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-0185; UL1TR002003 (NIH)
Record Dates: First submitted 2021-03-02; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Cerebral Blood Flow; Exercise
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — Exercise; histaminol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analysis assessor will be blinded to pre and post-testing samples, as well as to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training (EXT) (Active Comparator): Research participants will complete six weeks of supervised progressive aerobic and resistance exercise training (EXT). Cardiopulmonary, cerebral and peripheral vascular function will be measured pre and post EXT.
  Interventions: Other: Supervised Exercise Training Protocol
- Inspiratory Muscle and Exercise Training (IMET) (Experimental): Research participants will complete six weeks of supervised aerobic and resistance exercise training in addition to supervised respiratory muscle training (IMET). IMET sessions will be performed similar to EXT, with the exception of having sessions of at-home IMT training. On these days, all training will be spread out over a 2-hour session with periods of IMT training occurring at the beginning, middle, and end of the session. Cardiopulmonary, cerebral and peripheral vascular function will be measured pre and post IMET.
  Interventions: Other: Supervised Exercise Training Protocol; Other: Inspiratory Muscle and Exercise Training

INTERVENTIONS:
Other: Supervised Exercise Training Protocol — EXT: Supervised EXT will include a progressive individualized program that combines aerobic and resistance protocols. Volume progression will begin with 3-days of supervised training sessions/wk and will increase by 1 session/wk to a maximum of 5-days/wk. Each EXT session will include 30 minutes of aerobic training (15 minutes cycling; 15 minutes treadmill walking/running/elliptical) and 30 minutes of resistance training (specifics below). Considering individual fatigue will be a concern, therefore similar to exercise training standards in COPD, the duration of rest periods may be extended (~1-3 min) as needed, however, all exercise durations will be completed within a 1.5-hour time slot. On days that EXT and IMET interventions overlap, the training and IMET will be spread out over a 2-hour session as opposed to the 1.5-hour time slot.
  Other Names: EXT
Other: Inspiratory Muscle and Exercise Training — Inspiratory Muscle Training (IMT): All IMT sessions will be performed similar to EXT, with the exception of having 2-3-sessions of at-home IMT training depending on where in the exercise progression the individual is (i.e., Week1 vs week 6). On the days that IMT and exercise training overlap, all training will be spread out over a 2-hour session with periods of IMT training occurring at the beginning, middle and end of the session. Each week will include a measure of Maximal Inspiratory Pressure (MIP) and a Test of Inspiratory Respiratory Endurance (TIRE). The intensity of the IMT will be 50% of the weekly MIP, thus progressive increases in IMT threshold intensity will remain at 50% of the weekly MIP. In contrast, the TIRE protocol will assess respiratory endurance based on the relative baseline intensity. Thus TIRE testing will begin at a MIP intensity of 50% (weeks 1-2), and then progressing to 65% (weeks 3-4), and 80% (weeks 5-6).
  Other Names: IMET
  Arms: Inspiratory Muscle and Exercise Training (IMET)

SUMMARY:
Background: Respiratory and cardiovascular complications have emerged as dominant threats during and following coronavirus disease (COVID19) infection. Severe COVID19 infection is categorized as acute respiratory dysfunction leading to hospitalization, where as a mild infection is identified as symptoms of dyspnea, muscle pains, migraines, palpitations and/or fatigue persisting for several weeks. Recovery from COVID19 infection is poorly characterized, but symptoms appear to gradually decline over a four to eight-week period. Unfortunately, recovery from severe infection is similar to symptoms experienced with mild infection making it rather difficult to provide a physiological definition of recovery for mild infection sufferers. Considering that 81% of COVID19 infections are found to be mild, approximately 4.5 million Americans may be vulnerable to inadequate cardiovascular recovery that exacerbates reductions in physical capacity and quality of life. Combined respiratory muscle and exercise training enhance cardiorespiratory function, maximize return to activities of daily living, and reduces hospitalization times in heart failure, sepsis and severe acute respiratory syndrome. However, it is unclear if these interventions will also enhance cardiorespiratory and cerebrovascular COVID19 recovery. Therefore, utilizing cardiorespiratory and cerebrovascular rehabilitation techniques we propose these specific research aims and hypotheses to investigate the following:

1. Does individualized cardiac exercise rehabilitation enhance cardiorespiratory & cerebrovascular recovery?

   Hypotheses:
   1. Individualized exercise therapy designed to increase fitness will enhance cardiorespiratory function at rest, as well as during and following exercise in individuals recovering from COVID19.
   2. Cerebrovascular function at rest, as well as during and following exercise will be enhanced following individualized exercise therapy in individuals recovering from COVID19 infection.
   3. The magnitude of post-training cardiorespiratory enhancements will be associated with cerebrovascular adaptations in individuals recovering from COVID19 infection.
2. Does combining inspiratory muscle and cardiac exercise rehabilitation provide additive cardiorespiratory and cerebrovascular COVID19 recovery benefits?

Hypotheses:

1. The addition of inspiratory muscle training to individualized exercise therapy will enhance cardiorespiratory adaptation in individuals recovering from COVID19 infection.
2. Improved cardiorespiratory function associated with inspiratory muscle training and exercise therapy will add further recovery advantage to cerebrovascular function in individuals recovering from COVID19 infection.

Study Design Scientific Plan: This project aims to collect pre- and post-intervention cardiorespiratory and cerebrovascular measures in individuals 1- 4 weeks after recovering from COVID19 infection (n=40; 20 ♀ & 20♂). Each participant will be randomized to either Supervised Exercise Training (EXT; n=20) or combined inspiratory muscle and exercise testing (IMET; n=20) interventions. Randomization will match for age and sex, and will attempt balanced matching of any cardiovascular (hypertension, atherosclerosis), respiratory (chronic obstructive pulmonary disease, asthma), and metabolic (diabetes, metabolic syndrome) comorbidities between interventions. Prior to beginning EXT or IMET, participants will complete baseline fitness, respiratory muscle testing, cardiovascular, and cerebrovascular measures to DEXA body composition scan (dual energy X-ray absorptiometry, DEXA) determine the initial intensity and post-intervention effectiveness, respectively. Following baseline testing, participants will complete a 6-week EXT or IMET intervention. EXT: Supervised EXT will include a progressive individualized program that combines aerobic and resistance protocols. Volume progression will begin with 3-days of supervised training sessions/wk and will increase by 1 session/wk to a maximum of 5-days/wk. Each EXT session will include 30 minutes of aerobic training (15 minutes cycling; 15 minutes treadmill walking/running/elliptical) and 30 minutes of resistance training (specifics below). Considering individual fatigue will be a concern, therefore similar to exercise training standards in COPD, the duration of rest periods may be extended (~1-3 min) as needed, however all exercise durations will be completed within a 1.5-hour time slot. IMET: All IMET sessions will be performed similar to EXT, with the exception of having 3-sessions of at home IMT training. On these days, all training will be spread out over a 2-hour session with periods of IMT training occurring at the beginning, middle and end of the session.

DETAILED DESCRIPTION:
Aim 1 - Does individualized cardiac exercise rehabilitation enhance cardiorespiratory & cerebrovascular recovery? It is widely accepted that "exercise is medicine"; a polypill and a cornerstone in the prevention and recovery from disease, including those with similar pathogenicity to COVID19 (e.g., severe acute respiratory syndrome, middle eastern respiratory syndrome, and acute respiratory distress syndrome). More specifically, exercise is considered vascular medicine, capable of improving the vitality of arteries by healing the endothelium. Targeted, repeated, and episodic increases in blood flow and arterial shear stress during individualized bouts of exercise mechanically stimulate the endothelium, triggering the production of nitric oxide and other vasoactive and anti-inflammatory molecules required for vasculogenesis and angiogenesis. Therefore, exercise healing of the primary vascular structure that the SARS-CoV2 virus damages, provides significant regenerative vascular benefit to end organs like the lungs, heart, and brain. For instance, several cornerstone cardiorespiratory benefits derived from exercise therapy to treat various cardiorespiratory diseases are listed to highlight the feasibility of enhancing COVID19 recovery using individualized exercise interventions: 1) aerobic fitness is linked with attenuated endothelial dysfunction in the peripheral arteries following acute H1N1 infection; 2) restoration of lung elasticity and strength, as well as increased antioxidants that reduce inflammation following exercise training contributes to improving cardiorespiratory capacity; and 3) improved autonomic modulation of the cardiorespiratory system improves exercise capacity and overall health.

While there is minimal evidence that specifically demonstrates cerebrovascular function is altered following COVID19 infection, epidemiological evidence indicates individuals recovering from COVID19 have a higher risk of stroke. The earlier movement-based exercise rehabilitation is introduced for stroke treatment, the greater the improvement in exercise capacity, peripheral vascular and cerebrovascular function, largely because of attenuated vascular inflammation and increase neurotrophic modulators. Physical inactivity in individuals who have suffered a stroke or are at a high risk of stroke further exacerbates inflammatory vascular dysfunction. Exercise directly stimulates the cerebrovascular endothelium, by increasing blood flow and intra-arterial shear stress in cerebral arteries. Cerebrovascular function is regulated by an exquisite synergistic and redundant set of physiological controllers (i.e., arterial partial pressure of carbon dioxide and oxygen, arterial blood pressure, neurogenic autonomic modulation, and cardiac output). In addition to direct cerebrovascular benefits of exercise therapy, systemic cardiorespiratory improvements that enhance gas exchange, blood pressure, autonomic reflexes, and cardiac function will have important vascular benefits in the brain. Therefore, the proposed research provides significant benefit to improving exercise capacity, as well as cardiorespiratory and cerebrovascular function during recovery from COVID19 infection.

Cardiorespiratory function is quantified using a standardized battery of clinical tests to assess cardiovascular and pulmonary function at rest and during submaximal and maximal stressors. For instance, resting cardiovascular function is determined by measuring heart rate, left and right ventricular cardiac function, peripheral vascular blood flow, and pulse wave velocities. These metrics provide quantifiable information pertaining to arterial stiffness, autonomic and peripheral vascular function, which are primary determinants in regulating central hemodynamics (i.e., cardiac output, arterial blood pressure, and blood flow) and cardiovascular health. It is unknown if COVID19 infection impacts resting central hemodynamics. However, our research group has previously observed central hemodynamic dysfunction following acute inflammatory responses to different viral infections. Submaximal (flow mediated dilation) and maximal (cardiopulmonary exercise testing) physiological measures allow for researchers to quantify the cardiorespiratory systems ability to respond to stressors observed in daily activity. Following rehabilitation interventions, submaximal and maximal cardiopulmonary testing provides necessary quantification of the exercise interventions' effectiveness.

Cardiac Echocardiography: Left and right ventricular mechanics (end diastolic and end systolic volumes, mitral filling,), as well as central hemodynamics in the aorta and vena cave (aortic diameter, cardiac output, stroke volume, heart rate), will be assessed at rest using two-dimensional echocardiography via a Hitachi Aloka Alpha 7 system (Tokyo, Japan). With subjects in the left lateral position, measurements will be obtained using the two and four-chamber view. The interior of the left ventricle will be traced manually during both end systole and end diastole. Volumes will be measured using Simpson's rule. Stroke volume will be calculated by subtracting end diastolic volume from end systolic volume. Cardiac output will be calculated as HR multiplied by Stroke volume. Three beats will be measured, and the average will be used in the analyses. Ejection fraction will be calculated from the ventricular volumes and expressed as a percentage of end systolic to end diastolic volume. Mitral valve velocities will be obtained from the apical 4 chamber view, whereby E, A, and E/A will be measured. The slope of the inflow will also be determined. Tissue Doppler will also be performed to obtain E' with E/E' calculated. Lastly, speckle tracking will be performed using TOMTEC tissue tracking software.

Cerebrovascular function is traditionally assessed using a uni-dimensional approach, quantifying cerebral blood flow (CBF) responses to a single perturbation that stresses one of the primary mechanisms involved in CBF regulation. The primary mechanisms involved in CBF regulation at rest and during exercise are arterial blood gases, arterial blood pressure, neurogenic autonomic systems, and metabolism. Thus clinical stimuli are used to provoke a cerebrovascular response by altering environmental, pharmacological, or physiological conditions, that specifically perturb one of these primary mechanisms. Novel approaches, developed by our research team advance traditional uni-dimensional CBF assessments, by testing the cerebral vasculature using a battery of clinical assessments, or through assessments that evoke specific and systemic physiological perturbations that influence CBF. The two cerebrovascular assessment strategies utilized in this protocol specifically assess the cerebrovascular response to changes in carbon dioxide, blood pressure, and neurogenic activity at rest, as well as during incremental whole body and fatiguing hand grip exercise. These tests will provide traditional unidimensional quantification of cerebrovascular function, as well as providing nuanced quantification of integrative cerebrovascular function. Additionally, utilizing assessment strategies that similarly target the same systems that the training interventions aim to improve (i.e., respiratory, cardiovascular, and skeletal muscle systems), the pre and post intervention cerebrovascular tests will provide an index of the proportion that each system contributes to physiological recovery following our COVID19 infection.

Aim 2 - Does combining inspiratory muscle and cardiac exercise rehabilitation provide additive cardiorespiratory and cerebrovascular COVID19 recovery benefits? Pulmonary dysfunction and pneumonia are the predominant concerns of COVID19 infection. While fever, cough, fatigue, myalgia, and dyspnea are the most common symptoms in individuals infected by the COVID19 virus. For many individuals infected by COVID19, surviving the virus is only a portion of the problem. A recent report identified that COVID19 patients deemed to be recovered and thus discharged from hospital have a lingering abnormal pulmonary diffusion; a retrospective investigation revealed that pulmonary diffusion following COVID19 infection can remain abnormal for 30-days after discharge. Prolonged pulmonary impairment is primarily attributed to respiratory muscle atrophy and ventilator-induced diaphragm dysfunction in severe COVID19 infection. However, a prolonged bout of coughing, fatigue, and dyspnea associated with mild COVID19 infection can also trigger pulmonary dysfunction and impair respiratory muscle strength. Pulmonary dysfunction caused by poor inspiratory muscle strength increases work of breathing, muscle sympathetic nerve activity, and fatigue associated with physical activity. Fatiguing inspiratory muscle work reduces exercise and physical capacity, while increased muscle sympathetic nerve activity reduces blood flow to active limbs and increases fatigue. Consequently, lingering impairments in pulmonary function following COVID19 infection, regardless of severity, lowers exercise capacity, physical capabilities, quality of life, and likely cardio and cerebrovascular function.

Inspiratory muscle training, which effectively involves standardized breathing routines organized similar to exercise training programs, has proven effective at reducing fatigue, myalgia, and dyspnea in other chronic respiratory diseases. The improvement in cardiorespiratory function following IMT is primarily the result of strengthened inspiratory muscles. Elevating inspiratory muscle strength reduces the work of breathing during physical activity and metabolic cost associated with breathing both at rest and during physical activity. Skeletal muscles often compete for blood supply during exercise, especially when work of breathing is heightened, therefore improved inspiratory muscle function with IMT in conjunction with exercise training likely provides a hyper additive blood flow stimulus throughout the vasculature compared to exercise training alone. Considering the vasogenic and angiogenic properties derived from increased cardiovascular blood flow, IMT training in conjunction with exercise training provides an innovative strategy to facilitate an enhanced COVID19 recovery. No study to date has investigated the impact of IMT training and exercise on cerebrovascular function. However, improvements in cardiorespiratory function associated with improved respiratory muscle function should also synergistically enhance cerebrovascular regulation.

To summarize, the IPL specializes in utilizing exercise to improve the function of the cardiorespiratory and cerebrovascular systems in clinical models of chronic disease. For instance, members of the IPL have previously demonstrated that the cerebrovascular response to exercise, is dependent on carbon dioxide, arterial blood pressure, and arterial shear stress in health and disease. Moreover, individualized cardiac exercise rehabilitation increases CBF (~10%), re-establishing normal CBF, in heart failure populations. Similarly, the IPL has collected data related to the proposed research, in that exercise training improves vascular hemodynamics and autonomic modulation in populations living with inflammatory disease (diabetes); as well as improves blood pressure. The cardiorespiratory research specialists in the IPL have also demonstrated that muscle training improves exercise tolerance and dyspnea in obese patients who are at increased risk of complications from COVID infection. Collectively, researchers in the IPL aim to utilize these techniques and approaches to determine optimal strategies to enhance COVID19 recovery in the heart, brain, and lungs.

ELIGIBILITY:
Inclusion Criteria:

* BMI<40,
* 1-4 weeks post active COVID19 infection
* physician approval for undertaking exercise testing and training.
* Adequate intracranial ultrasound windows

Exclusion Criteria:

* Lingering COVID19 symptomology
* cardiovascular disease
* pulmonary disease
* cerebrovascular disease
* taking medication that influences heart rate, blood pressure, or cerebrovascular function,
* severe obesity (BMI >40)
* metabolic comorbidities (diabetes, metabolic syndrome),
* recently been diagnosed with a mild traumatic brain injury (within past 6 months).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Cerebrovascular Function | week 0 and week 7
  Change in cerebral artery vasodilatory capacity and stiffness using transcranial and vascular duplex ultrasound in individuals previously infected with COVID19 following six weeks of exercise training or exercise and inspiratory muscle training.
Cardiopulmonary Fitness | week 0 and week 7
  Change in cardiopulmonary fitness using incremental maximal exercise and measures of oxygen consumption in individuals previously infected with COVID19 following six weeks of exercise training or exercise and inspiratory muscle training.
Inspiratory Muscle Function | Week 1 and Week 6
  Change in inspiratory muscle function using tests of incremental respirayory endurance in individuals previously infected with COVID19 following six weeks of exercise training or exercise and inspiratory muscle training.

SECONDARY OUTCOMES:
Cerebrovascular metaboreflex | week 0 and week 7
  Change in cerebral artery metaboreflex using transcranial ultrasound in individuals previously infected with COVID19 following six weeks of exercise training or exercise and inspiratory muscle training.
Cardiac mechanics | week 0 and week 7
  Change in right and left ventricular mechanics using echosonography in individuals previously infected with COVID19 following six weeks of exercise training or exercise and inspiratory muscle training.
Peripheral artery function | Week 0 and 7
  Change in brachial and femoral artery endothelial function and arterial stiffness in individuals previously infected with COVID19 following six weeks of exercise training or exercise and inspiratory muscle training.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Smith, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided